CLINICAL TRIAL: NCT00244010
Title: Hematopoietic Stem Cell Transplantation (HSCT) From Partially Matched Family Donors for Patients With Refractory Severe Aplastic Anemia or Refractory Cytopenias: A Pilot Study
Brief Title: Partially Matched Stem Cell Transplantation for Patients With Refractory Severe Aplastic Anemia or Refractory Cytopenias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAAHAP; Severe Aplastic Anemia; Cytopenias
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2009-02

CONDITIONS: Anemia, Aplastic; Amegakaryocytic Thrombocytopenia; Diamond-Blackfan Anemia; Kostmann Syndrome
Keywords: Aplastic anemia; Amegakaryocytic thrombocytopenia; Diamond-Blackfan Anemia; Kostmann syndrome; Allogeneic stem cell transplantation; Haploidentical stem cell transplant; T-cell depletion; Partially matched family member donor transplant; Refractory cytopenia
MeSH Terms: conditions — Anemia, Aplastic; Anemia, Diamond-Blackfan; Neutropenia, Severe Congenital, Autosomal Recessive 3; Cytopenia | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Device: Allogeneic stem cell transplant

INTERVENTIONS:
Device: Allogeneic stem cell transplant — Participants will receive a reduced intensity conditioning regimen consisting of fludarabine, thiotepa, melphalan, and OKT3 followed by an infusion of haploidentical stem cells. Rituximab will be administered within 24 hours of the infusion in an effort to prevent posttransplant lymphoproliferative disorder LPD. In addition to T-cell depletion of the donor product, participant will receive mycophenolate mofetil for prophylaxis of GVHD.
  Other Names: Allogeneic stem cell transplantation; Haploidentical stem cell transplant; T-cell depletion; Partially matched family member donor transplant; Hematopoietic stem cell transplant

SUMMARY:
Due to an overall and disease free survival of 85% to 100%, allogeneic blood or bone marrow stem cell transplantation using an HLA matched sibling donor is the therapy of choice for patients with severe aplastic anemia (SAA). Unfortunately, only about 25% of patients have such a donor. For patients with SAA lacking a matched sibling donor, immunosuppressive therapy is the current treatment of choice. Approximately 70% of these patients have a complete or partial response to immunosuppressive therapy, achieving transfusion independence and/or growth factor independence.

For the approximately 30% of patients who do not respond to immunosuppressive therapy or experience recurrence, alternative donor (matched unrelated, partially matched family member) transplantation is a treatment option. However, graft rejection and graft-versus-host-disease (GVHD) are significant barriers to success, decreasing event-free survival to 30% to 50%.

This study offers stem cell transplantation using a partially matched family member (haploidentical) donor to those patients with no available HLA-matched sibling or matched unrelated donor. In an attempt to reduce GVHD and regimen-related toxicity while maintaining adequate engraftment, we plan to infuse a highly purified stem cell graft. The Miltenyi Biotec CliniMACS CD3 depletion system will be used to derive a defined allogeneic graft highly enriched for CD34+ hematopoietic cells and depleted of CD3+ T-lymphocytes from G-CSF mobilized, donor-derived peripheral blood stem cells.

Patients 21 years of age and younger with refractory cytopenias are also eligible for this protocol as there are no other potentially curative therapies currently available for these conditions.

The primary objective of this study is to evaluate the safety of transplantation using a haploidentical donor product engineered to targeted cell counts using the investigational CliniMACS device for patients with refractory severe aplastic anemia (SAA) or refractory cytopenias. The treatment plan would be considered unsafe if we can find this type of procedure is associated with a significantly higher treatment failure rate. Treatment failure is defined as any occurrence of the following events, overall grade III-IV acute GVHD, graft failure or death due to any cause within 100 days after transplant.

DETAILED DESCRIPTION:
Secondary objectives for this protocol include the following:

* To observe the degree of hematopoietic chimerism in T-cells during the first year posttransplant.
* To observe the relative proportions of donor/host T-regulatory cells during the first year posttransplant.
* To monitor rates of acute and chronic GVHD during the first year posttransplant.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:
* Refractory severe aplastic anemia
* Refractory Kostmann syndrome
* Refractory Diamond-Blackfan anemia
* Refractory amegakaryocytic thrombocytopenia
* Absence of a suitable HLA-matched sibling donor and absence of a 10/10 allele matched unrelated donor.
* Life expectancy of greater than six weeks as per the judgment of the principal investigator.
* Karnofsky or Lansky Performance Status score of greater than or equal to 70%.
* Creatinine clearance is greater than or equal to 40 cc/min/1.73 m2.
* FVC greater than or equal to 40% of predicted or pulse oximetry greater than or equal to 92% on room air.
* Does not have a known allergy to murine products.

Exclusion criteria:

* Ejection fraction or shortening fraction below the lower limit of normal for age.
* Lactating (female patient).
* Pregnant or lactating
* Diagnosis of Fanconi Anemia.
* Positive HLA crossmatch with donor

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kasow, DO, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two patients and two donors were enrolled between 10/24/2005 and 2/24/2009 when the study was closed. The study was terminated due to the PI leaving St. Jude.
Groups:
- Patients: Patients were enrolled to treat refractory severe aplastic anemia.
- Donors: Parents of patients were enrolled onto the SAAHAP study to provide hematopoietic stem cells.
Period: Overall Study
Arm/Group | Patients | Donors
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Donors | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failures
Description: The primary objective of this study is to evaluate the safety of HAPLO HSCT for patients with refractory severe aplastic anemia (SAA) or refractory cytopenias. The treatment plan would be considered unsafe if we can demonstrate that it is associated with a significantly higher treatment failure rate. The treatment failure is defined as any occurrence of the following events, overall grade III-IV acute GVHD, graft failure or death due to any cause within 100 days post HSCT or after the last cellular product infusion, if required.
Time Frame: 100 days post transplant
Population: Enrollment was terminated due to the PI leaving the institution. Insufficient data was generated to answer the objective.
Arm/Group | Patients | Donors
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Two patients and two donors were enrolled between 10/24/2005 and 2/24/2009 when the study was closed.
Groups:
- Donor: Donors were not assessed for adverse events.
Arm/Group | Patients | Donor
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=2) | Donor (N=0)
Cellulitis of skin (Infections and infestations) | 1 (1) | 0 (0)
Infection, Staphylococcus Aureus, Blood (Infections and infestations) | 1 (1) | 0 (0)
Methemoglobinemia (Investigations) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (intermittent) (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=2) | Donor (N=0)
Elevated Ferritin Level (Metabolism and nutrition disorders) | 1 (1) | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0
Fever without Neutropenia (General disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 1 (1) | 0
Hemosiderosis (Metabolism and nutrition disorders) | 1 (1) | 0
Hepatomegaly (intermittent) (Hepatobiliary disorders) | 1 (1) | 0
Nausea and Vomiting (intermittent) (Gastrointestinal disorders) | 1 (1) | 0
Pain-Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Iron overload (intermittent) (Metabolism and nutrition disorders) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
This study has terminated due to the PI leaving the institution. An insufficient number of subjects were enrolled to answer the primary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes